CLINICAL TRIAL: NCT06190834
Title: Relationship Between High Density Lipoprotein Subtypes and Prognosis in Coronary Heart Disease Patients.
Brief Title: Relationship Between High-Density Lipoprotein Subtypes and Coronary Heart Disease Prognosis.
Acronym: RHDLS-CHD
Status: Recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Guangdong Guosheng Medical Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-RHDLS-CHD
Record Dates: First submitted 2023-10-30; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-09

CONDITIONS: HDL; Coronary Heart Disease
Keywords: High-Density Lipoprotein; Subtypes; Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The patients with coronary heart disease diagnosed by coronary angiography: The patients with coronary heart disease diagnosed by coronary angiography in the department of cardiology of Beijing Tsinghua Changgeng Hospital. Except patients with severe valvular disease, severe myocarditis, severe hepatic and renal insufficiency, thyroid insufficiency, severe infectious or systemic inflammatory diseases, severe blood diseases, malignant tumors, etc.

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of human mortality worldwide, imposing substantial societal and economic burdens. Traditionally, high-density lipoprotein (HDL) has been branded as the "beneficial" lipoprotein. The Framingham study found that for every 1mg/dl increase in HDL, the risk of coronary heart disease (CHD) was reduced by 2% in men and 3% in women. Subsequent studies further affirmed the inverse correlation between HDL and the risk of CHD. However, these findings were first challenged by Mendelian randomization studies which failed to identify a causal relationship between HDL and CHD. Moreover, randomized controlled trials demonstrated that therapeutically increasing plasma HDL concentrations did not reduce the risk of CHD events, prompting doubts about HDL's status as "good cholesterol." The relationship between HDL and CHD might be more intricate than previously believed, possibly not just mediated by the quantity of HDL but also intimately linked with its function.

Several cross-sectional studies have confirmed the relationship between HDL subtypes and the severity of disease in CHD patients, yet findings are inconsistent. Conventional testing methods lack a universally accepted standard for defining or describing HDL subfractions, with issues like expensive equipment, poor repeatability, cumbersome operation, slow analysis, and low throughput. Microfluidic electrophoresis technology combines the merits of electrophoresis with microfluidic chip technology. This method facilitates efficient separation of substances in microchannels on a substrate, providing rapid and consistent results. Utilizing the latest microfluidic chip technology for HDL subfraction detection offers quick, accurate, and straightforward analysis with minimal sample volume and automation. It precisely reflects the serum concentrations of HDL subfractions HDL2b and HDL3, addressing the current pitfalls of clinical HDL subfraction analysis methods. This approach is poised to become the standard method for HDL subfraction testing.

In conclusion, existing studies on the association between HDL subtypes and CHD remain inconsistent, with most having a small sample size. Our study, leveraging microfluidic chip technology for HDL subfraction detection, aims to further investigate: the prognostic value of HDL subtypes for the long-term outcomes of CHD patients, building a risk prediction model for adverse cardiovascular events that includes HDL subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the patients is over 18 years old;
2. Coronary artery disease was confirmed by coronary angiography.

Exclusion Criteria:

1. Severe valvular disease, severe myocarditis, severe hepatic and renal insufficiency, thyroid insufficiency, severe infectious or systemic inflammatory diseases, severe blood diseases, malignant tumors.
2. Lack of data on HDL subtypes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with coronary heart disease diagnosed by coronary angiography in the department of cardiology of Beijing Tsinghua Changgeng Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of the major adverse cardiovascular event (MACE) | From date of enrollment until the date of first documented progression or date of MACE, whichever came first, assessed up to 3 years.
  MACE includes cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and planned coronary reconstruction therapy.
  Cardiovascular Death: Death due to cardiac causes, such as myocardial infarction, heart failure, arrhythmia, etc. Non-Fatal Myocardial Infarction: If a patient survives this condition, it is called a nonfatal myocardial infarction. Non-Fatal Stroke: A stroke is a neurological disorder caused by disruption of the blood supply to the brain. A non-fatal stroke means that the patient has experienced a stroke but survived. Unplanned Coronary Revascularization: This event refers to the unplanned reconstruction of the coronary arteries, which may involve either interventional therapy (such as coronary angioplasty) or surgical procedures (such as coronary artery bypass surgery).

SECONDARY OUTCOMES:
Number of the all-cause death | From date of enrollment until the date of first documented progression or date of all-cause death, whichever came first, assessed up to 3 years
  Deaths from all causes occurred between definitive diagnosis and the end of follow-up.
Number of the heart failure | From date of enrollment until the date of first documented progression or date of heart failure, whichever came first, assessed up to 3 years
  For patients who already have organic heart disease can not engage in any physical work, even in the state of rest, there are heart failure symptoms, which are significantly worse after a little activity.
In-stent restenosis | From date of enrollment until the date of first documented progression or date of in-stent restenosis, whichever came first, assessed up to 1 years
  In-stent restenosis is defined as an angiogram diameter stenosis of 50% or more in one segment of the stent or 5mm segment adjacent to the stent.
Number of the target lesion revascularization | From date of enrollment until the date of first documented progression or date of the target lesion revascularization, whichever came first, assessed up to 1 years.
  Target lesions include the 5mm range within the stent as well as the proximal and distal end of the stent. Repeated interventional therapy or bypass surgery for this segment is the target lesion revascularization.
Number of the non-target lesion revascularization | From date of enrollment until the date of first documented progression or date of the non-target lesion revascularization, whichever came first, assessed up to 1 years.
  Non-target lesion revascularization, including PCI or CABG, due to progression of the original lesion or newly formed lesions in areas other than the target lesion.
Number of the major adverse cardiovascular event (MACE) | From date of enrollment until the date of MACE during hospitalization.
  MACE includes cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and planned coronary reconstruction therapy.
Number of the major adverse cardiovascular event (MACE) | rom date of enrollment until the date of first documented progression or date of MACE, whichever came first, assessed up to 1 years.
  MACE includes cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and planned coronary reconstruction therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Geng, Study Director — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
undecided whether to share
Supporting Information: Study Protocol